CLINICAL TRIAL: NCT03879915
Title: Dental Implants in Patients With X-linked Hypophosphatemia
Acronym: IMPLANTS-XLH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: HAO 018045
Record Dates: First submitted 2019-03-15; First posted 2019-03-19 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: X-linked Hypophosphatemia
Keywords: hypophosphatemia; hypophosphatemic rickets; dental implants; osseointegration
MeSH Terms: conditions — Familial Hypophosphatemic Rickets; Hypophosphatemia; Rickets, Hypophosphatemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective Dental Implant placement: Patients prospectively included and treated following current recommendations
  Interventions: Procedure: Dental Implant placement
- Retrospective Dental Implant placement: Patients retrospectively included, that did not benefit from current recommendations
  Interventions: Procedure: Dental Implant placement

INTERVENTIONS:
Procedure: Dental Implant placement — Surgical placement of dental implant not associated with prior or concurrent bone augmentation

SUMMARY:
X-linked hypophosphatemia (XLH) is a rare genetic skeletal disease where increased phosphate wasting in the kidney leads to hypophosphatemia and prevents normal mineralization of bone and dentin, with osteomalacia as a principal manifestation. In previous works, the investigators have shown that adults with XLH present with more frequent and severe periodontitis than in the general population, and that vitamin D and phosphate supplementation improves their periodontal health, as it does for the osteomalacia. Their medical records also reveal that early implant failure is dramatically increased in these patients, when no supplementation is implemented, and standard surgical protocols followed. In contrast, the investigator's preliminary data showed that successful osseointegration was achieved with supplementation prior and after implant placement and extended healing time. Here, the investigators propose to assess the current recommendations for implant therapy in XLH patients, with 24 implants placed. The current recommendations consist of: 1) supplementation with vitamin D and phosphate for 3 months prior to implant placement and 6 months after; 2) implant healing time extended to 6 months. If osseointegration is achieved, prosthesis will be fabricated. Radiographic and clinical examination at 6, 12, 18 and 24 months after placement of the definitive restoration will evaluate the implant osseointegration, crestal bone level and peri-implant tissues health.

DETAILED DESCRIPTION:
Primary objective: to evaluate the efficacy of the specific implant management currently offered to XLH patients according to the recommendations, in terms of implant survival.

Secondary objectives: 1. to study the evolution of the peri-implant bone level within 2 years after implant placement ; 2. to study the evolution of the stability of the peri-implant tissues in the 2 years following the installation of the implant ; 3. to describe the osseointegration of the implant 6 months after insertion ; 4. to evaluate the effectiveness of the specific implant management in terms of the delay in occurrence of the first implant loss of patients ; 5. to describe the reasons for removal of the implants ; 6. to evaluate the satisfaction of the implant treated patient ; 7. to describe the occurrence of dental plaque, suppuration or bleeding around implants.

Experimental plan: this is an observational prospective study with historical control group (retrospective compendium) comparing XLH-specific implant management (prior phosphorus / vitamin D supplementation and prolonged implant healing) to non-specific management. For prospective inclusion (patients with specific implant management) patients will be recruited from adults with XLH as part of an oral assessment. After inclusion each patient will be followed 24 months. The surgical treatment and the clinical and radiographic follow-up correspond to the specific management proposed in our service to the patients presenting an XLH. Prior to implant placement, a cone-beam computed tomography scan will confirm adequate bone volume for implant placement. Implant surgery will be performed under local anesthesia following the protocols recommended by the manufacturer. The follow-up is done during the healing period and the realization of the implant prosthesis (6 months after surgery) then 12, 18 and 24 months after the surgery. It will include a clinical and radiographic examination, and will verify the presence of the implant in the mouth (survival of the implant), and the stability of the peri-implant tissues (level of attachment and bone level)

ELIGIBILITY:
Prospective patients:

Inclusion criteria

* Man or woman
* 18 years of age or older at the time of inclusion
* Diagnosis of X-linked hypophosphatemia confirmed by an endocrinologist or a rheumatologist
* Supplemented with phosphate and vitamin D for a period of at least 3 months
* Presenting an indication of a simple implant treatment (healed implant site with adequate bone volume) with rehabilitation using a single or partial fixed prosthesis
* Affiliated to the national social security assurance

Exclusion Criteria:

* Opposition to participation in research
* Presence of other uncontrolled diseases that may have an impact on the periodontium (eg diabetes or chronic kidney disease)
* Contraindications to implant treatment, such as active periodontitis and heavy smoking (more than 10 cigarettes per day)
* Patient under guardianship or trusteeship.

Retrospective control patients:

The data will be collected retrospectively for patients who meet the following criteria:

* Man or woman
* Aged 18 years or older at the time of implant treatment
* Diagnosis of X-linked hypophosphatemia confirmed by an endocrinologist or a rheumatologist
* Having had non-specific XLH implant treatment (absence of phosphate / vitamin D supplementation and / or absence of prolonged healing)
* Non opposition to the use of the data of care collected as part of the research
* Absence at the time of implant treatment of uncontrolled diseases that may have had an impact on the periodontium (diabetes, chronic kidney disease, smoking > 10 cigarettes per day)
* Not under guardianship or trusteeship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with X-linked hypophosphatemia
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2019-09-27 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Implant loss | 24 months
  Loss of the dental implant within 24 months after placement, defined by the absence of the implant in the mouth objectified during a clinical examination (spontaneous loss) or by the removal of the implant whatever the cause

SECONDARY OUTCOMES:
Peri-implant bone level | 24 months
  Peri-implant bone level measured on dental x-rays
Clinical attachment level | 24 months
  Clinical attachment level, calculated from the pocket depth and gingival level measures and measured with a periodontal probe
Lack of mobility of the implant | 6 months
  Lack of mobility of the implant
Time of onset of the first implant loss | 24 months
  Time of onset of the first implant loss
Cause of removal of the implant | 24 months
  Cause of removal of the implant
Satisfaction of the treated patient | 24 months
  Satisfaction (or not) of the treated patient
Presence of dental plaque, suppuration or bleeding at the level of the implant | 24 months
  Presence of dental plaque, suppuration or bleeding at the level of the implant

CONTACTS AND LOCATIONS:
Overall Officials: Martin Biosse Duplan, DDS, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service d'Odontologie - Hôpital Bretonneau - 23 rue Joseph de Maistre, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided